CLINICAL TRIAL: NCT03531879
Title: ARROW: identificAtion of postpRandial biomaRkers tOWards Cardiovascular Prevention
Brief Title: ARROW:identificAtion of postpRandial biomaRkers tOWards Cardiovascular Prevention
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: Institute for Human Development and Potential (IHDP), Singapore (Other); National Heart Centre Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 17.15.NRC
Record Dates: First submitted 2018-05-09; First posted 2018-05-22 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- subject with plaques and without plaques: Subject with plaques and without plaques

SUMMARY:
The purpose of this study is to better understand the association between the postprandial biomarker responses after a food challenge with the development of cardiovascular diseases in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to sign written informed consent in English or Chinese prior to trial entry
2. 40-54 years old
3. Both male and female subjects
4. Chinese ethnic group (having both grandparents Chinese)
5. Low Framingham risk of CHD (<10%)
6. Apparently healthy (i.e. no chronic or ongoing acute disease), based on investigator's clinical judgement

Exclusion Criteria:

1. Food allergy to any of the constituents of the meal challenge (milk proteins, lactose, soy).
2. Subjects not willing or not able to comply with scheduled visits and the requirements of the study protocol.
3. Contraindication to MRI
4. Pregnant or lactating women based on investigator's clinical judgement.
5. Morbid obesity (BMI ≥ 40 kg/m2).
6. Previous myocardial infarction (MI). This will include ST-elevation MI (STEMI) and non-ST-elevation MI (NSTEMI).
7. Known coronary artery disease - prior coronary revascularization.
8. Known documented peripheral arterial disease.
9. Previous stroke (defined as new focal neurological deficit persisting more than 24hours).
10. Use of anti-hypertensive agents.
11. Prior history of cancer (excludes pre-cancerous lesions).
12. Life expectancy less than 1 year.
13. Known definite diabetes mellitus or on treatment for diabetes mellitus.
14. Known autoimmune disease or genetic disease.
15. Known endocrine and metabolic diseases, even on treatment, including hyperlipidemia.
16. Psychiatric illness.
17. Asthma or chronic lung disease requiring long term medications or oxygen.
18. Chronic infective disease, including tuberculosis, hepatitis B and C; and HIV.
19. Currently participating or having participated in another clinical trial within 4 weeks prior to trial start (except for Biobank Study and SingHeart).

Ages: 40 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study will be performed in 100 Chinese subjects at low risk of developing cardiovascular diseases, as defined by the Framingham Heart Study Coronary Heart Disease 10-year risk score with or without subclinical atherosclerosis.
Sampling Method: Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2019-06-14 (Actual)

PRIMARY OUTCOMES:
To compare the kinetics of postprandial biomarkers between two groups of healthy subjects with and without subclinical atherosclerosis | Within 28 days from enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Nestle Research Center, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Loh X, Sun L, Allen JC, Goh HJ, Kong SC, Huang W, Ding C, Bosco N, Egli L, Actis-Goretta L, Magkos F, Arigoni F, Yeo KK, Leow MK. Gender differences in fasting and postprandial metabolic traits predictive of subclinical atherosclerosis in an asymptomatic Chinese population. Sci Rep. 2022 Oct 7;12(1):16890. doi: 10.1038/s41598-022-20714-6. PMID 36207366
- [Derived] Valsesia A, Egli L, Bosco N, Magkos F, Kong SC, Sun L, Goh HJ, Weiting H, Arigoni F, Leow MK, Yeo KK, Actis-Goretta L. Clinical- and omics-based models of subclinical atherosclerosis in healthy Chinese adults: a cross-sectional exploratory study. Am J Clin Nutr. 2021 Nov 8;114(5):1752-1762. doi: 10.1093/ajcn/nqab269. PMID 34476468